CLINICAL TRIAL: NCT02652988
Title: Home-based Transcranial Direct Current Stimulation in Fibromyalgia Patients. Phase II, Randomized, Double-blind, Single-center Clinical Trial
Brief Title: Home-based Transcranial Direct Current Stimulation in Fibromyalgia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wolnei Caumo (Other)
Responsible Party: Sponsor-Investigator, Wolnei Caumo, Wolnei Caumo, DIRECTOR OF PAIN&NEUROMODULATION LAB, Hospital de Clinicas de Porto Alegre
Organization: Hospital de Clinicas de Porto Alegre (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-0471
Record Dates: First submitted 2015-10-28; First posted 2016-01-12 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Fibromyalgia
Keywords: tDCS; chronic pain; fibromyalgia
MeSH Terms: conditions — Fibromyalgia; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active-tDCs (Active Comparator): 17 patients will receive Active-tDCS intervention (2mA, 30 min) at home.
  Interventions: Other: Active-tDCS
- Sham-tDCS (Sham Comparator): 17 patients will receive Sham-tDCS intervention (2mA, 30 min) at home.
  Interventions: Other: Sham-tDCS

INTERVENTIONS:
Other: Active-tDCS — Active home-based tDCS applied at home.
  Arms: Active-tDCs
Other: Sham-tDCS — Sham home-based tDCS applied at home.
  Arms: Sham-tDCS

SUMMARY:
In this phase II, randomized, double-blind clinical trial, the investigators intended to evaluate the home-based effect of transcranial direct current stimulation (tDCS) in patients with fibromyalgia. This syndrome affects between 3-5% of the population in an age group 40-60 years also occurring in childhood and old age. Reaches 3.4% of women and 0.5% of men. Fibromyalgia is a chronic widespread pain syndrome in various parts of the body. The neuromodulation techniques have as a principle produce inhibition or cortical arousal. The tDCS is a non-invasive brain stimulation method used to modulate the cortical excitability, using a low intensity direct current (1-2mA) directed to the scalp via the cathode and anode electrodes. The current reaches the cortex, producing hyperpolarization or depolarization of the axonal membrane potential. Evidence has shown that this method is presented as a technique able to alter cortical and subcortical neural networks. This technique has been used to treat psychiatric disorders such as depression, acute mania, bipolar affective disorder, panic, hallucinations, obsessive compulsive disorder, schizophrenia, withdrawal, rehabilitation after stroke, pain syndromes such as neuropathic pain, migraine, pancreatitis pain chronic and fibromyalgia. The tDCS is a low cost technique, with virtually no side effects and which exerts therapeutic effect by neuromodulatory pathways by distinct pathways activated by the drugs. In this scenario falls within the importance of developing this device for home use by fibromyalgia patients, since it is easy to use and thereby enables maintaining the benefit observed in studies performed and supervised frequently used in care centers. The use of tDCS over the long term is not feasible in hospital by patients demands, sometimes every day or more than once a week, removing the patient from their activities, and cost shifting and overload the healthcare system. Therefore, the objective of this study is to evaluate the effect of home-based tDCS in fibromyalgia patients in long-term treatment.

DETAILED DESCRIPTION:
Will be included women aged between 18 and 65 years, chronic pain fibromyalgia according to the criteria of the American College of Rheumatology, pain unresponsive to analgesics such as paracetamol, acetylsalicylic acid, ibuprofen, Carisoprodol, Zanaflex (Tizanidine) and Codeine. And give informed consent to participate after initial evaluation. Primary outcome is to evaluate the effect of treatment with home-base tDCS in patients with fibromyalgia. Secondary outcomes are: compare the effect of active home-based tDCS and sham in cortical neurophysiological processes and subcortical to stimulation with TMS and standardized noxious stimuli with and without concomitant conditioned Pain Modulation (CPM) in pain threshold outcomes to the test mechanical pressure, heat-algesic stimulus, cortical excitability parameters [evoked rest motor (MEP) MEP enough to evoke amplitude of 1 mV peak to peak, silent period (SP), motor threshold (MT), variation in blood volume and oxygenation cortical motor area [oxy-hemoglobin concentrations (Hbo) / deoxy-hemoglobin (HBr)] optically functional neuroimaging (NIRS) and variation in the frequency of alpha and beta waves of motor area stimulated by tDCS assessed by electroencephalogram (EEG). In surrogate outcome, the investigators will compare the effect of active home-sham tDCS the tDCS in pain levels and functional capacity, catastrophic thinking, bookmark levels of neurotrophic activity (BDNF) and astrocytic (S100 beta).

ELIGIBILITY:
Inclusion Criteria:

* have chronic pain fibromyalgia according to the criteria of the American College of Rheumatology
* Pain unresponsive to analgesics such as paracetamol, acetyl salicylic acid, Ibuprofen, Carisoprodol, Zanaflex (Tizanidine) and Codeine
* Give informed consent to participate after initial evaluation.

Exclusion Criteria:

* Pregnancy
* Treatment with carbamazepine and gabapentin
* The. Metallic implant in the brain
* Medical devices implanted in the brain
* Alcohol or drug abuse history in the last 6 months
* Suffering from severe depression (with score> 30 on the Beck Depression Inventory)
* History of neurological disorders
* Unexplained fainting History
* History of head trauma or momentary loss of consciousness (self reported)
* Neurosurgery History
* Decompensated systemic diseases, and chronic inflammatory diseases (lupus, rheumatoid arthritis, renal failure and hepatitis).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01; Primary Completion 2018-05-01 (Actual); Study Completion 2018-06-12 (Actual)

PRIMARY OUTCOMES:
Pain level in fibromyalgia patients using home-based tDCS | Ffive days per week, during 12 weeks.
  Evaluate the level of pain in fibromyalgia patients before and after each home-based tDCS session. We will use numerical pain scale to do that.

SECONDARY OUTCOMES:
Serum levels of Brain Derived Neurotrophic Factor (BDNF) | 2 days
  Measurement of serum levels of BDNF pre and pos application of home-based application of home-based tDCS
Serum levels of calcium-binding protein B (S100B) | 2 days
  Measurement of serum levels of S100B pre and pos application of home-based tDCS
Functional capacity | 2 days
  Measurement of functional capacity pre and pos application of home-based tDCS with functional capacity scale in chronic pain.
Catastrophic thinking | 2 days
  Measurement of catastrophic thinking pre and pos application of home-based tDCS with catastrophizing scale.

CONTACTS AND LOCATIONS:
Overall Officials: Wolnei S Calmo, Ph.D, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (2):
- Brazil (2):
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Wolnei Caumo, Porto Alegre, Rio Grande do Sul

REFERENCES:
- [Background] Arnold LM. Biology and therapy of fibromyalgia. New therapies in fibromyalgia. Arthritis Res Ther. 2006;8(4):212. doi: 10.1186/ar1971. PMID 16762044
- [Background] Ablin J, Fitzcharles MA, Buskila D, Shir Y, Sommer C, Hauser W. Treatment of fibromyalgia syndrome: recommendations of recent evidence-based interdisciplinary guidelines with special emphasis on complementary and alternative therapies. Evid Based Complement Alternat Med. 2013;2013:485272. doi: 10.1155/2013/485272. Epub 2013 Nov 21. PMID 24348701
- [Background] Bigatti SM, Hernandez AM, Cronan TA, Rand KL. Sleep disturbances in fibromyalgia syndrome: relationship to pain and depression. Arthritis Rheum. 2008 Jul 15;59(7):961-7. doi: 10.1002/art.23828. PMID 18576297
- [Background] Boggio PS, Rigonatti SP, Ribeiro RB, Myczkowski ML, Nitsche MA, Pascual-Leone A, Fregni F. A randomized, double-blind clinical trial on the efficacy of cortical direct current stimulation for the treatment of major depression. Int J Neuropsychopharmacol. 2008 Mar;11(2):249-54. doi: 10.1017/S1461145707007833. Epub 2007 Jun 11. PMID 17559710
- [Background] Bradley LA, Wohlreich MM, Wang F, Gaynor PJ, Robinson MJ, D'Souza DN, Mease PJ. Pain response profile of patients with fibromyalgia treated with duloxetine. Clin J Pain. 2010 Jul-Aug;26(6):498-504. doi: 10.1097/AJP.0b013e3181dee80e. PMID 20551724
- [Background] Bymaster FP, Dreshfield-Ahmad LJ, Threlkeld PG, Shaw JL, Thompson L, Nelson DL, Hemrick-Luecke SK, Wong DT. Comparative affinity of duloxetine and venlafaxine for serotonin and norepinephrine transporters in vitro and in vivo, human serotonin receptor subtypes, and other neuronal receptors. Neuropsychopharmacology. 2001 Dec;25(6):871-80. doi: 10.1016/S0893-133X(01)00298-6. PMID 11750180
- [Background] Burgmer M, Pogatzki-Zahn E, Gaubitz M, Wessoleck E, Heuft G, Pfleiderer B. Altered brain activity during pain processing in fibromyalgia. Neuroimage. 2009 Jan 15;44(2):502-8. doi: 10.1016/j.neuroimage.2008.09.008. Epub 2008 Sep 24. PMID 18848998
- [Background] Clauw DJ. Fibromyalgia: an overview. Am J Med. 2009 Dec;122(12 Suppl):S3-S13. doi: 10.1016/j.amjmed.2009.09.006. PMID 19962494
- [Background] Chappell AS, Bradley LA, Wiltse C, Detke MJ, D'Souza DN, Spaeth M. A six-month double-blind, placebo-controlled, randomized clinical trial of duloxetine for the treatment of fibromyalgia. Int J Gen Med. 2008 Nov 30;1:91-102. doi: 10.2147/ijgm.s3979. PMID 20428412
- [Background] Chen R, Samii A, Canos M, Wassermann EM, Hallett M. Effects of phenytoin on cortical excitability in humans. Neurology. 1997 Sep;49(3):881-3. doi: 10.1212/wnl.49.3.881. PMID 9305361
- [Background] Fregni F, Gimenes R, Valle AC, Ferreira MJ, Rocha RR, Natalle L, Bravo R, Rigonatti SP, Freedman SD, Nitsche MA, Pascual-Leone A, Boggio PS. A randomized, sham-controlled, proof of principle study of transcranial direct current stimulation for the treatment of pain in fibromyalgia. Arthritis Rheum. 2006 Dec;54(12):3988-98. doi: 10.1002/art.22195. PMID 17133529
- [Background] Fregni F, Boggio PS, Nitsche MA, Marcolin MA, Rigonatti SP, Pascual-Leone A. Treatment of major depression with transcranial direct current stimulation. Bipolar Disord. 2006 Apr;8(2):203-4. doi: 10.1111/j.1399-5618.2006.00291.x. No abstract available. PMID 16542193
- [Background] Fregni F, Boggio PS, Nitsche M, Pascual-Leone A. Transcranial direct current stimulation. Br J Psychiatry. 2005 May;186:446-7. doi: 10.1192/bjp.186.5.446. No abstract available. PMID 15863752
- [Background] Giesecke T, Williams DA, Harris RE, Cupps TR, Tian X, Tian TX, Gracely RH, Clauw DJ. Subgrouping of fibromyalgia patients on the basis of pressure-pain thresholds and psychological factors. Arthritis Rheum. 2003 Oct;48(10):2916-22. doi: 10.1002/art.11272. PMID 14558098
- [Background] Harris RE, Clauw DJ. Newer treatments for fibromyalgia syndrome. Ther Clin Risk Manag. 2008 Dec;4(6):1331-42. doi: 10.2147/tcrm.s3396. PMID 19337439
- [Background] Lindell L, Bergman S, Petersson IF, Jacobsson LT, Herrstrom P. Prevalence of fibromyalgia and chronic widespread pain. Scand J Prim Health Care. 2000 Sep;18(3):149-53. doi: 10.1080/028134300453340. PMID 11097099
- [Background] Manganotti P, Bongiovanni LG, Zanette G, Turazzini M, Fiaschi A. Cortical excitability in patients after loading doses of lamotrigine: a study with magnetic brain stimulation. Epilepsia. 1999 Mar;40(3):316-21. doi: 10.1111/j.1528-1157.1999.tb00711.x. PMID 10080512
- [Background] Mease P. Fibromyalgia syndrome: review of clinical presentation, pathogenesis, outcome measures, and treatment. J Rheumatol Suppl. 2005 Aug;75:6-21. PMID 16078356
- [Background] Moore RA, Cai N, Skljarevski V, Tolle TR. Duloxetine use in chronic painful conditions--individual patient data responder analysis. Eur J Pain. 2014 Jan;18(1):67-75. doi: 10.1002/j.1532-2149.2013.00341.x. Epub 2013 Jun 3. PMID 23733529
- [Background] Roizenblatt S, Fregni F, Gimenez R, Wetzel T, Rigonatti SP, Tufik S, Boggio PS, Valle AC. Site-specific effects of transcranial direct current stimulation on sleep and pain in fibromyalgia: a randomized, sham-controlled study. Pain Pract. 2007 Dec;7(4):297-306. doi: 10.1111/j.1533-2500.2007.00152.x. Epub 2007 Nov 6. PMID 17986164
- [Background] Schestatsky P, Stefani LC, Sanches PR, Silva Junior DP, Torres IL, Dall-Agnol L, Balbinot LF, Caumo W. Validation of a Brazilian quantitative sensory testing (QST) device for the diagnosis of small fiber neuropathies. Arq Neuropsiquiatr. 2011 Dec;69(6):943-8. doi: 10.1590/s0004-282x2011000700019. PMID 22297885
- [Background] Staud R. Treatment of fibromyalgia and its symptoms. Expert Opin Pharmacother. 2007 Aug;8(11):1629-42. doi: 10.1517/14656566.8.11.1629. PMID 17685881
- [Background] Staud R, Smitherman ML. Peripheral and central sensitization in fibromyalgia: pathogenetic role. Curr Pain Headache Rep. 2002 Aug;6(4):259-66. doi: 10.1007/s11916-002-0046-1. PMID 12095460
- [Background] Valle A, Roizenblatt S, Botte S, Zaghi S, Riberto M, Tufik S, Boggio PS, Fregni F. Efficacy of anodal transcranial direct current stimulation (tDCS) for the treatment of fibromyalgia: results of a randomized, sham-controlled longitudinal clinical trial. J Pain Manag. 2009;2(3):353-361. PMID 21170277